CLINICAL TRIAL: NCT00498732
Title: Dissection of Differentially Expressed Genes and Pathways in Patients With Obstructive Sleep Apnea Syndrome Before and After CPAP Treatment
Brief Title: Dissection of Differentially Expressed Genes and Pathways in Patients With OSAS Before and After CPAP Treatment
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Peilin Lee/Attending physician, National Taiwan University Hospital
Other Study IDs: 200701064R
Record Dates: First submitted 2007-07-08; First posted 2007-07-10 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive sleep apnea syndrome; CPAP, microarray
MeSH Terms: conditions — Sleep Apnea, Obstructive; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CPAP — CPAP treatment for 4 weeks

SUMMARY:
Specific Aim

1. To verify the differentially expressed genes and pathways between normal and OSA patients, and OSA patients before and after CPAP treatment.

   Genes with changes in expression of more than two-fold between normal and OSA patients as well as OSA patients before and after CPAP treatment were thought as confirmed and were selected for further validation study.
2. To correlate the confirmed genes with the clinical presentations and CPAP effects in another 50 OSAS subjects to validate the altered gene expressions and pathways involved.

   To investigate the correlation of genes confirmed from RT-PCR (identified gene), another 50 OSAS subjects are included in the study. We analyze the correlation between identified gene and the clinical manifestations and CPAP effect in these 50 OSAS patients.
3. To establish a cell model to investigate the differentially expressed genes and the putative biological pathways involved in OSA syndrome.

To investigate the functions of genes identified in the first and second year (gene of interest), we establish a cell model with human monocyte cell line U937. We investigate the function of gene of interest through overexpress or knockdown.

Objectives The objectives of this project are to confirm the gene profiled from comparing normal and OSA patients as well as OSA patients before and after CPAP treatment, to investigate the correlation between altered gene expression and clinical presentations and CPAP effects of the OSAS and to identify and confirm corresponding pathway. This study will enhance our understanding of the individual constitution on widely different clinical characteristics and therapeutic variations. All these efforts will also help us to interpret its molecular mechanisms and develop prediction and diagnosis strategies of OSAS. The long-term objectives are to develop therapeutic strategy other than CPAP of OSAS.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is characterized with recurrent collapse of upper airway during sleep and resulted in hypoxia and sleep fragmentation, which resulted in cardiovascular diseases, metabolic disorders and neurocognitive dysfunctions. The cardiovascular complications attributed to OSAS included hypertension, coronary artery disease, heart failure and stroke. The mechanisms responsible for developments of cardiovascular sequelae included repeated episodes of hypoxia and hypercapnia, exaggerated negative intrathoracic pressure and bursts of sympathetic activity provoking surges in blood pressure and heart rate. Increase of inflammatory mediators, which included C-reactive protein, oxidative stress, adhesion molecules, vascular endothelial growth factor and proinflammatory cytokines, were thought to involve in the developments of cardiovascular diseases in patients with OSAS.

To clarify the exact mechanisms of OSAS and the linkage to cardiovascular complications, in our previous study, we used oligo microarray to genome-wide profile the gene expression patterns in OSAS patients and the changes of gene expressions before and after four-week CPAP treatment. The oligo-microarray data were processed with CRSD database and two-way hierarchical clustering method. The results showed the gene expression patterns were different between control subjects and OSA patients and CPAP treatment also altered the gene expression patterns. Totally 27 genes and four pathways were identified as target genes and pathways from comparing the gene pattern changes before and after CPAP treatment, which included apoptosis, oxidative phosphorylation, cell adhesion and activation and metabolism. To continue analyzing the gene pattern changes before and after CPAP treatment, we propose this three-year project to achieve the following goals: (1) To verify the differentially expressed genes and pathways between normal and OSA patients, and OSA patients before and after CPAP treatment. (2) To correlate the confirmed genes with the clinical presentations and CPAP effects in another 50 OSAS subjects to validate the altered gene expressions and pathways involved. (3) To establish a cell model to investigate the differentially expressed genes and the putative biological pathways involved in OSA syndrome. The information obtained by this approach is very useful to understand the pathogenic mechanism of OSA that leads to systemic complications and further therapeutic intervention may therefore be possible.

ELIGIBILITY:
Inclusion Criteria:

* Severe obstructive sleep apnea (AHI>=30/hr) age, sex, BMI match control subject

Exclusion Criteria:

* Refused to participate in this study
* Had severe obstructive pulmonary disease or active neurological events
* Enrolled in other studies at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From patients who were referred to sleep lab for suspect sleep apnea, we selected 50 male patients with age> 18 y/o. with severe OSAS, which were confirmed with by overnight PSG. All were free from neurologic events, chronic pulmonary disease, active infection and substance abuse. Female patients and patients under 18 y/o were excluded. All 50 subjects were treated with 4-week CPAP. All study subjects were admitted, on the day of baseline measurement and four weeks after CPAP use, for clinical evaluation, blood sampling and PSG. And all anti-hypertensive therapy was remained unchanged during the 4-week follow-up period. Changes of parameters, before and after CPAP treatment, were compared between two groups.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-03 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peilin Lee, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan